CLINICAL TRIAL: NCT06943950
Title: A Randomized, Double-blind, Placebo-controlled Phase III Study to Evaluate the Efficacy and Safety of SYHX1901 Tablets in the Treatment of Moderate to Severe Plaque Psoriasis
Brief Title: A Phase III Study of SYHX1901 Tablets in the Treatment of Moderate to Severe Plaque Psoriasis
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SYHX1902-007
Record Dates: First submitted 2025-04-17; First posted 2025-04-25 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Moderate to Severe Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SYHX1901 dose 1 (Experimental)
  Interventions: Drug: SYHX1901
- SYHX1901 dose 2 (Experimental)
  Interventions: Drug: SYHX1901
- Placebo (Placebo Comparator)
  Interventions: Drug: SYHX1901

INTERVENTIONS:
Drug: SYHX1901 — Administered orally, once daily (QD)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of different doses of SYHX1901 tablets in the treatment of moderate to severe plaque psoriasis.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled phase III study to evaluate the efficacy and safety of three different doses of SYHX1901 tablets compared with placebo in the treatment of moderate to severe plaque psoriasis. The total duration of the study will be 60 weeks which will be comprised of: a screening period (4 weeks); a core treatment period (16 weeks), a extended treatment period（36 weeks）and a follow-up assessment period (4 weeks). Eligible subjects will be randomly assigned to SYHX1901 dose 1 , dose 2 or placebo group at a 2:2:1 ratio for continuous oral administration for 16 weeks，then placebo group will will be randomly assigned to SYHX1901 dose 1, dose 2 at a 1:1 ratio for continuous oral administration for 36 weeks, the SYHX1901 dose 1, dose 2 group will remain the same dose for 36 weeks. The presence or absence of prior treatment with biological agents will be a stratification factor. Subjects will be monitored for the efficacy and safety throughout the study.

ELIGIBILITY:
Inclusion Criteria:

Subjects fully understand and voluntarily participate in this study and sign informed consent; 2. Age ≥18 and ≤ 65 years old; 3. Subjects with a clinical diagnosis of stable moderate-to-severe plaque psoriasis with a history ≥6 months before randomization; Subjects with stable moderate-to-severe plaque psoriasis defined as meeting all four of the following criteria simultaneously:

1. Subject must be diagnosed of chronic plaque psoriasis with no morphological changes or significant outbreaks of disease activity assessed by the investigator;
2. Subject must be a candidate for systemic treatment or phototherapy assessed by the investigator;
3. Body Surface Area (BSA) affected by plaque-type psoriasis ≥10% at screening and baseline;
4. PASI score of ≥10 and Static Physician's Global Assessment (sPGA) score ≥3 at screening and baseline; 4. Negative blood pregnancy results should be provided 7 days (inclusive) prior to randomization, and subjects and their partners should voluntarily take contraceptive measures considered effective by the investigator during the study period and for at least 28 days after the study; 5. Subjects must be volunteer and be able to complete study procedures and follow-up examinations.

Exclusion Criteria:

1. Forms of psoriasis other than plaque psoriasis (Guttate psoriasis、erythrodermic psoriasis、Pustular psoriasis、Drug-induced psoriasis);
2. Previous or current autoimmune disease that may affect the clinical evaluation of psoriasis;
3. Other active skin conditions that may affect the clinical evaluation of psoriasis;
4. Active bacterial, viral, fungal, or other infection that requires medical intervention;
5. With progressive or uncontrolled systemic disease, or with chronic disease identified by the investigator as inappropriate for participation in the study;
6. History of malignancy ;
7. Any other medical and/or social reasons identified by the investigator as inappropriate for participation in the study;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-04-28 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Title: The Number of Participants With a Static Physician's Global Assessment (sPGA) Score of 0 or 1 in Participants Receiving SYHX1901 Compared to Placebo at Week 16 (sPGA 0/1) Description: The sPGA is a 5-point scale of an average assessment of all | Week 16
Title: The Number of Participants Who Achieve a 75% Improvement From Baseline in the Psoriasis Area and Severity Index (PASI) Score in Participants Receiving SYHX1901 Compared to Placebo at Week 16 (PASI 75) Description: PASI is a measure of th | Baseline and Week 16